CLINICAL TRIAL: NCT04999449
Title: Nebulizer Delivery of Intranasal Scopolamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jay C. Buckey Jr., Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001115
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Scopolamine; Motion Sickness
Keywords: Scopolamine; Motion Sickness; Space Physiology
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic study followed by double-blind, placebo-controlled, dose-ranging design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacokinetic (Experimental): Participants receive 1 dose of Scopolamine 0.4 mg delivered via a intranasal nebulizer developed by Creare LLC.
  Interventions: Drug: Scopolamine
- Chair (Experimental): Participants receive 1 dose of Scopolamine 0.2 mg, 1 dose of Scopolamine 0.4 mg, and 1 dose of placebo saline delivered via the Creare LLC intranasal nebulizer. These dosages are all 1 week apart and the order is randomized.
  Interventions: Drug: Scopolamine; Drug: Placebo

INTERVENTIONS:
Drug: Scopolamine — Intranasal scopolamine at 0.2 mg or 0.4 mg
Drug: Placebo — Intranasal saline placebo
  Arms: Chair

SUMMARY:
To develop a better way to administer anti-motion sickness medications using an intranasal nebulizer.

DETAILED DESCRIPTION:
An aqueous scopolamine formulation is being administered via a nebulizer and the pharmacokinetics of the drug are being measured.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Adults age 21-49
* Normal weight for body size, based on BMI table
* General good health, as determined by a verbally provided medical history
* Normal brief neurological exam
* Renal and hepatic function within normal ranges
* Able to provide written informed consent to participate

Exclusion Criteria:

* Drug allergies to scopolamine or other belladonna alkaloid
* Use of medications within 1 week of starting the study
* Use of an investigational drug within 30 days of starting the study
* Tobacco smoking within the past year
* Blood donation or significant blood loss within 30 days of starting the study
* Significant gastrointestinal disorder (e.g. Crohn's Disease, ulcerative colitis, chronic constipation), asthma, glaucoma, prostate problems, urinary obstruction, or seizure disorders
* History of alcohol or other drug abuse
* Pregnancy or suspected pregnancy, or lactation (pregnancy will be confirmed with urine pregnancy testing prior to drug administration)
* Consumption of grapefruit juice within 7 days of scopolamine (SCOP) administration
* Nasal, nasal sinus, or nasal mucosa surgery within 90 days prior to study initiation
* Other significant surgeries within 90 days
* Significant deviated septum that blocks air flow in one nostril
* Rhinitis, sinus infection, severe allergies, and other upper respiratory infections within 30 days prior to the study
* Current use of an intranasal medication
* Wheezing or other respiratory problem
* Unable to consent
* Prisoner

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Time to maximal concentration for scopolamine after intranasal administration (Tmax) | Baseline, 180 minutes
  Plasma scopolamine concentrations will be measured using an liquid chromatography-mass spectrometry (LC- MS) assay. Tmax is measured in minutes to reach the maximum concentration.
Side effects of intranasal scopolamine, as measured through a questionnaire with a subjective rating scale | 180 minutes
  A questionnaire will be administered asking about the participant's side effect profile after taking intranasal scopolamine. The questionnaire will have a subjective rating scale of 0-10 on the potential scopolamine side effects expected

SECONDARY OUTCOMES:
Effectiveness in reducing motion sickness as measured by duration of chair ride. | Baseline, end of chair ride (maximum of 20 minutes)
  The degree of motion sickness will be assessed by measuring the total number of minutes the subject rides in the chair before stopping

CONTACTS AND LOCATIONS:
Overall Officials: Jay C Buckey, Ph.D, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No